CLINICAL TRIAL: NCT07147621
Title: Evaluation of Chemotherapy-induced Cognitive Disorders During the Treatment of Hematological Malignancies
Acronym: HematoBrain
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0247
Record Dates: First submitted 2025-08-05; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patient group
- control group

SUMMARY:
Chemotherapy-induced cognitive disorders, such as memory problems, slowness of execution, inability to concentrate, and language difficulties, are sequelae that occur in patients undergoing chemotherapy or who have received chemotherapy. These symptoms lead to a degradation of the patients' quality of life and can have a significant social and familial impact. They are most commonly described in solid oncology, particularly in patients with breast cancer. Data about patients with hematological malignancies are scarce, but they seem to show the same phenomenon as in solid oncology. Indeed, many chemotherapies are used both in hematology and solid oncology and may therefore cause similar effects on cognition. Additionally, due to their mechanism of action, some chemotherapies specifically used in hematology could induce cognitive disorders. Hematology-treated patients are probably also affected by these disorders and may consequently experience a reduced quality of life.

The objective of this study is to assess the changes in cognitive functions in patients receiving chemotherapy for the treatment of hematological malignancies, using neuropsychological tests and a self-administered questionnaire, compared to a control group, as well as their potential impact on quality of life, fatigue, anxiety, and depression.

ELIGIBILITY:
Inclusion Criteria:

* Patient group inclusion criteria:

  * adult patient with acute myeloid leukemia, Hodgkin's lymphoma, or non-Hodgkin's lymphoma;
  * patient receiving a fixed-duration first-line chemotherapy;
  * patient affiliated or beneficiary of a social security scheme; .signed inform consent form.
* Control group inclusion criteria:

  * adult;
  * patient's relative (spouse, brother, sister, friend, etc.);
  * less than 5 years of difference with the patient;
  * same educational level (< baccalaureate/high school degree, baccalaureate/high school degree level, 2-year university degree, > 2-year university degree);
  * person affiliated or beneficiary of a social security scheme;
  * signed informed consent form

Exclusion Criteria:

* Patient group exclusion criteria:

  * no patient's relative for the control group;
  * known or suspective cognitive disorders prior to chemotherapy;
  * history of severe neurological or psychiatric disorders (e.g., severe depression); .previous chemotherapy;
  * previous brain radiotherapy;
  * ongoing treatments affecting cognition;
  * patient unable to read;
  * patient not speaking French;
  * person deprived of liberty by judicial or administrative decision;
  * person under forced psychiatric care;
  * person under legal protection measures;
  * person unable to express consent; .pregnant or breastfeeding woman.
* Control group exclusion criteria:

  * known or suspected cognitive disorders;
  * history of severe neurological or psychiatric disorder (e.g., severe depression); .previous chemotherapy;
  * previous brain radiotherapy;
  * ongoing treatments affecting cognition;
  * person unable to read;
  * person not speaking French;
  * person deprived of liberty by judicial or administrative decision;
  * person under forced psychiatric care;
  * person under legal protection measures;
  * person unable to express consent;
  * pregnant or breastfeeding woman."

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in the patient group will be recruited from the Hematology Departments of 2 French academic centers (Angers and Brest University Hospitals).
  Participants in the control group will be selected among the patient's relatives (family, friends, colleagues, etc.) of the same age category (less than 5 years of difference) and with the same education level.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Changes in cognitive complaints measured by the Functional Assessment of Cancer Therapy - Cognitive function (FACT-Cog) questionnaire | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  "Changes in cognitive complaints are measured by comparing the FACT-Cog scores obtained in the patient group and in the control group (intra- and inter-group comparison) before chemotherapy and 6 months after chemotherapy.
  The FACT-Cog questionnaire is a self-administered questionnaire used to measure cognitive complaints in cancer patients. It consists of 37 questions divided into 4 sections: Perceived Cognitive Impairment (20 questions, score range: 0-72), Comments From Others (4 questions, score range: 0-16), Perceived Cognitive Abilities (9 questions, score -range: 0-28), and Impact on Quality of Life (4 questions, score range: 0-16). Each question is assessed on a 5-point Likert scale. Higher scores indicate lower cognitive complaints."

SECONDARY OUTCOMES:
Changes in the scores obtained on the MoCA test | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the MoCA test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the WAIS-IV Information test | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the WAIS-IV Information test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the Hopkins Verbal Learning Test. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the Hopkins Verbal Learning Test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the TMT parts A and B. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the TMT parts A and B in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the WAIS-IV Codes test. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the WAIS-IV Codes test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the forward and reverse digit span memory test. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the forward and reverse digit span memory test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the Baddeley's dual task. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the Baddeley's dual task in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the 'P' and 'Animal' verbal fluency test. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the 'P' and 'Animal' verbal fluency test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the Stroop test. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the Stroop test in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy
Changes in the scores obtained on the quality of life questionnaire | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the EORTC QLQ-C30 (European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire for Cancer) in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the fatigue questionnaire. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the FACIT-Fatigue (Functional Assessment of Chronic Illness Therapy - Fatigue Scale) questionnaire in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Changes in the scores obtained on the anxiety and depression questionnaire. | Baseline At the end of the last chemotherapy cycle (up to 6 months after baseline, depending on the type of chemotherapy) Six months after chemotherapy (up to 1 year after baseline)
  Comparison of the scores obtained on the Hospital Anxiety and Depression Scale (HAD scale) in the patient group and in the control group before chemotherapy, after chemotherapy and 6 months after chemotherapy.
Logistic regression between patient's characteristics and evolution of cognitive complaints measured by the FACT-Cog questionnaire. | 6 months after chemotherapy
a) Correlation between the score on the FACT-Cog and the scores on objective neuropsychological tests (MoCA, WAIS-IV, Hopkins Verbal Test, WAIS-IV, TMT parts A and B, digit span memory test, Baddeley's dual, "P" and "Animal" verbal fluencies, stroop) | 6 months after chemotherapy
b) Correlation between the score on the FACT-Cog questionnaire and the scores on quality of life (EORTC-QLQ-C30), fatigue (FACIT-Fatigue), anxiety and depression (HADS) questionnaires | 6 months after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Angers, Angers, Maine et Loire, France